CLINICAL TRIAL: NCT06822387
Title: Growing an Extension Network for Multisite Dissemination and Implementation of Intensive Health Behavior and Lifestyle Treatment
Brief Title: Health Without Barriers/Salud Sin Barreras- Northern Colorado
Acronym: HWB/SSB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: Colorado State University Extension-Larimer County (Unknown); Colorado State University Extension-Weld County (Unknown); Colorado State University Extension-La Plata County (Unknown); University of Colorado, Denver (Other); United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5952
Record Dates: First submitted 2024-11-04; First posted 2025-02-12 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Lifestyle Risk Reduction; Adolescent Health; Family Health; Cardio-metabolic Health; Mental Health; Wellness Program; Type 2 Diabetes; Obesity, Adolescent
Keywords: Whole-family; Mindfulness; Wellness education; Nutrition; Physical Activity; Stress reduction; Health Without Barriers; Salud Sin Barreras
MeSH Terms: conditions — Risk Reduction Behavior; Psychological Well-Being; Diabetes Mellitus, Type 2; Pediatric Obesity; Motor Activity | interventions — Exercise; Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health without Barriers/ Salud Sin Barreras (HWB/SSB) (Experimental): HWB/SSB is a community-delivered, whole-family intensive health behavior and lifestyle intervention intended to reduce adolescent risk of chronic diseases (i.e., T2D) through promoting health behaviors and healthy stress management. The program is based on a lifestyle intervention called the Healthy Living Program (HeLP), a family-centered obesity prevention and treatment program for children. Previous and ongoing work has focused on tailoring HWB/SSB implementation to ensure cultural suitability for adolescents and their families in Southwest Colorado.
  HWB/SSB emphasizes "whole family" involvement including the participation of siblings, elders, other caregivers, and relatives. HWB/SSB is delivered.
  The HWB/SSB intervention delivery is not considered human subjects research; only the evaluation, dissemination, and implementation elements are considered research. The intervention will be delivered regardless of any research activity.
  Interventions: Behavioral: Mindfulness-Based Intervention; Behavioral: Parent Education; Behavioral: Physical Activity; Behavioral: Brief Mindfulness Intervention for Parents; Behavioral: Preschool Curriculum; Behavioral: Nutrition and Cooking Education

INTERVENTIONS:
Behavioral: Mindfulness-Based Intervention — Learning to BREATHE (L2B) is an evidence-based mindfulness curriculum for adolescents. L2B in this program consists of 6 sessions of approximately 1 hour per session. In between sessions, participants are asked to practice brief mindfulness skills individually.
Behavioral: Parent Education — The parent education curriculum includes 3 modules: 1) family support/parenting, 2) nutrition education and 3) physical activity education. Parents set weekly goals to implement what they learned in each session at home with their family.
Behavioral: Physical Activity — Focuses on using cardio and resistance training to improve cardiorespiratory health in youth.
Behavioral: Brief Mindfulness Intervention for Parents — Parent-based mindfulness education is based on the Learning to BREATHE curriculum.
Behavioral: Preschool Curriculum — Preschool age children learn about and try new foods.
Behavioral: Nutrition and Cooking Education — Nutrition education and hands-on cooking lessons for the whole family.

SUMMARY:
The overarching goal of this work is to address the limited access to evidence-based health behavior and lifestyle interventions for youth and families most impacted by preventable chronic diseases, including obesity and type 2 diabetes. In the current project, we implement a small single-arm pilot and feasibility trial of Health Without Barriers/Salud Sin Barreras (HWB/SSB), a culturally-adapted, whole-family intensive health behavior and lifestyle intervention to 11-19-year-old adolescents and their families living in Northern Colorado. Objectives are refining the HWB/SSB community facilitator training, evaluating the feasibility and acceptability of HWB/SSB implementation, and characterizing changes in health outcomes among adolescent participants.

DETAILED DESCRIPTION:
Health Without Barriers/Salud Sin Barreras (HWB/SSB) is a 12-session community-delivered, whole-family intensive health behavior and lifestyle intervention for health promotion and reduction of risk for chronic diseases (e.g., type 2 diabetes). The program is delivered over 6 weeks and includes mindfulness-based stress reduction training for adolescents, parent/caregiver health education and mindfulness training, youth physical activity, and whole-family nutrition education and cooking/meal preparation. Previous and ongoing work has focused on gathering and using direct input from local community members and families from Southwest Colorado to adapt HWB/SSB to ensure cultural suitability for teenagers and their families in this region. Now, there is a need for further refinement of HWB/SSB community facilitator training and evaluation of the intervention. The HWB/SSB intervention delivery is NOT considered human subjects research; only the evaluation, dissemination, and implementation elements are considered research (objectives described below). The intervention will be delivered regardless of any research study, and participation in the research study is not a requirement for families to enroll in HWB/SSB or for facilitators to facilitate the intervention.

There are three main objectives to this study:

1. Train community-based facilitators for HWB/SSB and refine training through: (a) conducting a series of focus groups with facilitators (up to n=20), (b) facilitator completion of a knowledge tests before and after training, (c) facilitator completion of surveys to evaluate and refine training processes, and (d) monitoring fidelity of HWB delivery through completion of standardized checklists by HWB trainers of mock and live sessions and through facilitator fidelity surveys.
2. Enroll adolescents (up to n=60) and parents/caregivers (up to n=60) from Northern Colorado in HWB/SSB to evaluate the acceptability and feasibility of the program. Program acceptability will be assessed through a series of focus groups and acceptability surveys completed by the participants. Program attendance and retention will be used to assess feasibility.
3. Describe changes in adolescents' psychological, health behavior, and health-related outcomes from before to up to 1-year after HWB/SSB participation. Outcomes include: 1) cardiometabolic health, 2) stress management, 3) enjoyment, self-efficacy, and frequency of physical activity, 4) healthy eating behaviors, and 5) sleep health.

ELIGIBILITY:
Inclusion Criteria:

Adolescent subjects

* Between the ages 11-19 years old
* Reside in Larimer County, Weld County, or the surrounding areas.

Parent/guardian subjects:

* 18 years old or older
* Are parents/guardians of an adolescent between the ages of 11-19
* Reside in Larimer County, Weld County, or the surrounding areas

Facilitators subjects

* 18 years old or older
* Reside in Larimer County, Weld County, or the surrounding areas
* Are planning to or have facilitated HWB

Exclusion Criteria

Adolescents subjects will not take part in the research activities if they have a medical and/or psychological/behavioral condition that, in the opinion of the Colorado State University/Extension program team, could interfere with safety for themselves or others or interfere with the capability of the participant or other participants to potentially benefit from the program (e.g., severe emotional-behavioral disturbance, inability to follow facilitator directions).

Parents/guardians will not take part in the research activities if they have a medical and/or psychological/behavioral condition that, in the opinion of the Colorado State University/Extension program team, could interfere with safety for themselves or others or interfere with the capability of their family or other participating families to potentially benefit from the program (e.g., using drugs or alcohol or under the use of drugs/alcohol during program sessions, aggressive or inappropriate behavior toward other participants).

There is no exclusion for facilitator subjects.

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Intervention Fidelity: Observer Session Ratings | 6 weeks
  HWB delivery fidelity will be assessed as percentage adherence to the curriculum, determined by HWB trainers ratings of HWB sessions on a standardized checklist. The range is 0% (no adherence) to 100% (complete adherence), with higher scores reflecting better adherence
Intervention Fidelity: Facilitator Session Ratings | 6 weeks
  HWB delivery fidelity will be assessed as percentage adherence to the curriculum, determined by HWB facilitator ratings of HWB sessions on a standardized checklist. The range is 0% (no adherence) to 100% (complete adherence), with higher scores reflecting better adherence
Intervention Acceptability: Questionnaire | 6 weeks
  Participants rate and comment on each component of the program (i.e. parent education, physical fitness, mindfulness, etc.) separately. Participants are asked to report on how supported they felt during the program, the helpfulness of the facilitators, the perceived benefits of program participation, and their overall experience participating in the program. This questionnaire will only be completed one time at the post-program follow-up. Intervention acceptability ratings can range from 1=not at all to 5=extremely, with higher scores reflecting better acceptability.
Intervention Feasibility: Attendance | 6 weeks
  Intervention feasibility will be assessed as percentage of family attendance of HWB sessions. The range is 0% (no attendance) to 100% (complete attendance), with higher scores reflecting better feasibility.

SECONDARY OUTCOMES:
Intervention Acceptability: Qualitative Themes | 6 weeks
  Adolescents and parents will participate in focus groups post-intervention to discuss their overall experiences with the program and its components. The discussion will explore aspects that were beneficial, identify challenges, and highlight areas for improvement. Themes related to the acceptability of the intervention will be derived from the qualitative analysis of the focus groups.
Intervention Training Evaluation: Qualitative Themes | 6 months
  Facilitators will participate in focus groups to discuss their experiences with the training and facilitation process, including aspects that were beneficial, challenges or areas for improvement, their confidence in facilitating, and their experiences working with families. Themes related to the evaluation of the intervention will be derived from the qualitative analysis of the focus group discussions
Intervention Training Fidelity: Facilitator Knowledge | 6 months
  Facilitators will complete knowledge test following the completion of the facilitator training. The purpose of these tests is to assess their understanding and retention of key concepts, skills, and principles that facilitators need to effectively deliver the intervention. The range is 0% to 100% with 100% reflecting better training.
Intervention Training Evaluation: Questionnaire | 6 months
  Facilitators will rate and comment on the training process of the HWB program. Questions include topics about how supported facilitators felt during the training process, previous experience in facilitating group programs, confidence in facilitating after the training, and feedback on any recommended modifications to training procedures that they perceive would improve the training process.
Emotional Regulation | 1 year
  Difficulties in Emotion Regulation Scale-Short Form (18 items), measures non-acceptance of emotional responses, difficulty engaging in goal-directed behavior, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity. Items are rated on a 5-point scale that range from 1 ("Almost never") to 5 ("Almost always"). Items are summed to calculate both a total score and subscale scores for each of the six domains. Higher scores are more negative, suggesting a greater degree of emotional dysregulation.
Positive Youth Development | 1 year
  Positive Youth Development- Very Short Form, measures positive indicators of child well-being including competence, confidence, character, connection, and caring. This measures has 17 items which are responded to on a 5-point scale ranging from 1 ("Strongly disagree") to 5 ("Strongly agree"). Items are averaged to calculate both a total score and subscale scores for each domains. High scores in each domain indicate stronger, more positive perceptions or experiences of positive development in that area, and higher overall scores suggest a higher level of positive youth development across all domains.
Dispositional Mindfulness | 1 year
  Mindful Attention Awareness Scale (MAAS) measures an individual's present-moment attention in daily living (dispositional mindfulness). The MAAS has 15 items which are responded to on a 6-point scale ranging from 0 ("Almost always") to 6 ("Almost never"). Items are averaged to calculate a total score. Higher scores reflect higher levels of dispositional mindfulness.
Eating behavior | 1 year
  Reward-Based Eating Drive Scale (REDS), a reliable/valid survey instrument of hedonic eating (reward-based eating). The RED has 13 items which are responded to on a 5-point scale ranging from 0 ("Strongly Disagree") to 4 ("Strongly agree). Scores are summed to calculate a total score. Higher scores indicate to greater propensity for reward-related eating.
Physical activity-engagement | 1 year
  NIH Patient-Reported Outcomes Measurement Information System (PROMIS): Pediatric Physical Activity - Short Form, measures the number of times an individual engaged in different types of physical activity in the past 7 days. This form has 4 items which are responded to on a 5-point scale ranging from 1 ("No days") to 5 ("6-7 days"). Items are summed to calculate a total score. Higher scores indicate more frequent engagement in physical activity.
Physical activity- self-confidence | 1 year
  Exercise Self-Efficacy Scale, measures an individual's beliefs in their ability to continue exercising on a three time per week basis at moderate intensities for 40 or more minutes per session in the future. This measure has 8 items which are responded to on a 100-point percentage scale comprised of 10-point increments, ranging from 0% ("not at all confident") to 100% ("highly confident"). The total self-efficacy score is calculated by summing the confidence ratings for all items and dividing by the total number of items in the scale. This produces a score with a maximum possible value of 100, where higher scores indicate greater exercise self-confidence.
Sleep Quality | 1 year
  Pittsburgh Sleep Quality Index, self-rated questionnaire that assesses sleep quality and disturbances over a 1-month interval. The PSQI has 19 self-rated questions. The 19 self-rated items are used to calculate seven "component" scores, each ranging from 0 to 3 points. A score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are summed to generate a single "global" score, with a range from 0 to 21 points. A score of "0" indicates no difficulties, while a score of "21" reflects severe difficulties across all areas. Higher scores indicate lower (poorer) sleep quality.
Cardiometabolic health: Lipid profile and HbA1c | 1 year
  Finger prick by lancet is used to analyze HbA1c, HDL/LDL cholesterol, and triglycerides.
Daily glucose patterns | 1 year
  Continuous glucose monitoring is used to describe average daily glucose, peak glucose, standard deviation, and mean amplitude of glycemic excursions.
Blood pressure | 1 year
  Blood pressure is assessed via digital blood pressure monitor.
Height | 1 year
  Height will be measured in centimeters using a stadiometer during the in-person research visits. Height and weight will be combined to report a both non-fasted and fasted BMI in kg/m^2.
Weight | 1 year
  Weight will be measured in using a calibrated scale at the in-person research visits. A fasting weight (10-hour overnight fast) using a smart scale for participants who opt-into this research activity. Weight and height will be combined to report both a non-fasted and fasted BMI in kg/m^2.
Body fat percentage | 1 year
  Body fat percentage is measured using bioelectrical impedance analysis (BIA).
Activity Monitoring | 1 year
  Participants will be fitted with a ActiGraph wGT3X-BT and asked to wear the device for 7 days.
Sleep Monitoring | 1 year
  Participants will be fitted with a ActiGraph wGT3X-BT and asked to wear the device for 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren B Shomaker, PhD, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No